CLINICAL TRIAL: NCT01586507
Title: A Single Dose Pharmacokinetic, Tolerability, and Safety Study of ULTRAM ER at Two Dose Levels in Adolescents Twelve to Seventeen Years Old, Inclusive, With Pain
Brief Title: A Study of ULTRAM ER at Two Dose Levels in Adolescents With Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR014017; TRAMAPPAI1003 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Pain
Keywords: Pain; ULTRAM ER; Tramadol hydrochloride; Adolescents
MeSH Terms: conditions — Pain | interventions — Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: ULTRAM ER
- Group 2 (Experimental)
  Interventions: Drug: ULTRAM ER

INTERVENTIONS:
Drug: ULTRAM ER — One dose of ULTRAM ER that is closest to 2 mg/kg, based on the participant's body weight and adjusting the dose in 25 mg increments.
  Arms: Group 1
Drug: ULTRAM ER — The target dose for Group 2 will be the one that achieves a level of exposure similar to that seen with a single 200 mg ULTRAM ER dose in adults.
  Arms: Group 2

SUMMARY:
The purpose of this study is to compare the pharmacokinetic (PK) of single oral doses of ULTRAM Extended Release (ER) at 2 dose levels in adolescents between 12 and 17 years old, inclusive (up to 17 years 364 days) with pain due to injury or nonmalignant disease, to the PK in adults, with respect to the PK parameter AUC∞ (area under the curve) of racemic tramadol. PK explores how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time.

DETAILED DESCRIPTION:
This is a multicenter, open-label (all people know the identity of the intervention), 2-group, single dose study. Within each group of participants for Parts 1 and 2, at least 1/3 of the participants will be female, at least 1/3 of the participants will be male, at least 1/3 of the participants will be below the age of 14 years, and at least 1/3 of the participants will be above the age of 16 years. Participants will be assigned to 1 group only. Each group of participants will receive a single oral dose of ULTRAM ER on 1 occasion. Group 1 will receive a dose of ULTRAM ER that is closest to 2 mg/kg, based on the participant's body weight and adjusting the dose in 25 mg increments. Following completion of all evaluations of Group 1, the pharmacokinetic data will be evaluated to target a dose for Group 2 that will achieve a level of exposure similar to that seen with a single 200 mg ULTRAM ER dose in adults. The maximum dose of ULTRAM ER should not exceed 6 mg/kg or 300 mg. When the study physician, the investigators, and the medical monitors agree that the PK of the drug is well-characterized and that the drug is well tolerated, enrollment will begin for Group 2 of the study. The sponsor's responsible Medical Officer will evaluate the safety of the calculated dose in Group 2 participants by evaluation of adverse drug events paying particular attention to events suggestive of either opioid toxicity or serotonin toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed need for control of pain due to injury or nonmalignant disease that does not influence fluid shifts and general drug disposition
* Weighs at least 30 kg
* Female participants must be premenarchal, surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control
* Able to swallow the intact tablet with the aid of water (participants may not chew, divide, dissolve, or crush the study drug)
* Signed informed consent document indicating that he/she understands the purpose of and procedures required for the study and is willing to participate in the study
* Informed consent signed by the parent(s) or the legal guardian(s) of the participant

Exclusion Criteria:

* History of or current clinically significant medical illness or condition including (but not limited to) cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness or condition that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The area under the curve (AUC∞) of ULTRAM ER as the primary PK parameter | At 1, 4, 6, 8, 12, 16, 24, 36, and 48 hours post dose

SECONDARY OUTCOMES:
Plasma concentration profile of ULTRAM ER | At 1, 4, 6, 8, 12, 16, 24, 36, and 48 hours post dose
Plasma concentration profiles of M1 and M5 metabolites | At 1, 4, 6, 8, 12, 16, 24, 36, and 48 hours post dose
Incidence of adverse events as a measure of safety and tolerability | 48 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Single Dose Pharmacokinetic, Tolerability, and Safety Study of ULTRAM ER at Two Dose Levels in Adolescents Twelve to Seventeen Years Old, Inclusive, with Pain — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2077&filename=CR014017_CSR.pdf